CLINICAL TRIAL: NCT06382740
Title: Prospective Evaluation of a Selection Protocol for Patients Over 70 Years Old for Liver Transplantation
Brief Title: Selection Protocol for Liver Transplantation in Patients Aged Over 70 Years
Acronym: Over70-LT
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Director, Azienda Ospedaliera di Padova
Other Study IDs: AOP2097
Record Dates: First submitted 2023-03-09; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: End Stage Liver DIsease; Liver Transplantation; Old Age
Keywords: liver transplantation; old recipients; age>70 years
MeSH Terms: conditions — End Stage Liver Disease | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Liver transplantation — Liver transplantation

SUMMARY:
Increased life expectancy and aging population has led to a trend of increasing liver transplant (LT) volume in the elderly. Nowadays, advanced age is not considered an absolute contraindication for LT but elderly LT candidates typically have an age-associated burden of comorbid conditions that can pose several clinical challenges during the selection/evaluation process for LT. Specific algorithms for elderly patient selection for LT are not well established; however, consensus agreement is that elderly LT candidates need a more rigorous selection process.

This study proposes a "step by step" algorithm of selection for liver transplant candidates more than 70 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >70 years and ≤ 75 years
* Liver transplant from cadaveric donor
* First liver transplant
* End stage liver disease or liver tumor

Exclusion Criteria:

* Age ≤ 70 years
* Living donor liver transplant
* Previous liver transplant
* Liver transplant for acute liver failure

Ages: 71 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Consecutive candidates for liver transplant with age >70 and ≤ 75 years
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
1 year patient survival | 12 months
  Overall patients survival at 12 months from liver transplantation

SECONDARY OUTCOMES:
1 year graft survival | 12 months
  Overall graft survival at 12 months from liver transplantation
3 months mortality and morbidity | 3 months
  Mortality and morbidity rates at 3 months from liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Cillo, Prof, Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- U.O.C Chirurgia Epatobiliare e Trapianti Epatici, Azienda Ospedaliera di Padova, Padua, Italy